CLINICAL TRIAL: NCT05551533
Title: Design and Pilot-test of an Innovative Mobile-based Intervention to Promote Mental Health of Informal Dementia Caregivers Through User-Centered Design
Brief Title: Mobile App Intervention for Informal Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Yuan Qi, Senior Research Fellow, Institute of Mental Health, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHG20.P.I.2.6
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Caregiver Burden; Dementia; Digital Health
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): To use the mobile app developed by the study team for one month. The app has a few key features including a positive reflection journal, online peer support, knowledge sharing, self-assessment, and locally available resources. Participants in the intervention group will be required to complete at least two positive reflection journal entries per week, and will be encouraged to use other features of the app during the one month period.
  Interventions: Other: Kampung Care App
- Wait list (No Intervention): Participants in this group will be put on a wait-list for one month before they can use the app.

INTERVENTIONS:
Other: Kampung Care App — Please refer to the previous session
  Arms: Intervention

SUMMARY:
Informal caregivers of persons with dementia (PWD) usually experience elevated levels of caregiving burden and potential depression. This project aims to develop and pilot-test a mobile app intervention for informal caregivers of PWD in Singapore. The project will have three phases in total including 1) phase 1 - to develop the app prototype and collect feedback from caregivers via focused group discussions. 2) a pilot RCT with 60 participants in total - 30 will be required to use the app for one month while another 30 will be on a waiting list for one month. and 3) in-depth interviews to seek users' feedback on the app for its future improvements. We hypothesize that the mobile app designed through a user-centered process would lead to high acceptance and high user engagement among local dementia caregivers. The 1-month intervention using the app developed subsequently would lower the reported depressive symptoms among local dementia caregiver. It will also improve their knowledge of dementia, caregiving efficacy, positive coping strategy, perceived positive aspects of caregiver and social support, and their mental well-being; and reduce their caregiving burden, and level of anxiety, compared to the control group.

DETAILED DESCRIPTION:
The prevalence of dementia was found to be 10% among residents aged 60 years and above in Singapore according to the Well-being of the Singapore Elderly study, equivalent to 51,934 older adults. As the population is aging in Singapore, and the fact that the incidence of dementia doubles with every 6.3-year increase in age after 60 years old, this number is going to grow as well, together with an increasing number of their informal caregivers. Informal caregivers of persons with dementia (PWD) usually experience elevated levels of caregiving burden from supporting the daily functioning of the PWD as well as issues such as work-family-caregiving conflicts and social isolation. These stressors can lead to potential depression among informal caregivers. The aggregate prevalence of depression was reported to be 34% according to a previous meta-analysis. Due to their heavy involvement in daily caregiving, caregivers usually have difficulties in attending face-to-face interventions. For instance, the average weekly hours spent on caregiving were reported to be 55 hours in our recent study among local informal caregivers. And this situation might be even worse in the current COVID-19 outbreak. To better support them now and in the future, an alternative could be to rely on a mobile-based intervention, as the penetration rate of smartphones among local residents is quite high (aged 15-49: >95%, aged 50-59: 88%, and aged 60 and above: 56%). Several studies have strengthened the evidence that these methods are feasible and acceptable among dementia caregivers. And preliminary evidence also suggested that such interventions were viable and potentially effective in promoting the mental health status among informal dementia caregivers.

This study aims to address the following gaps - Firstly, there is a lack of user-centered design in app development as well as rigorously designed studies based on a clear theoretical framework for dementia caregivers. Secondly, none of the existing evidence-based mobile apps for supporting dementia caregivers is Singapore-based. Lastly, a mobile-based intervention developed with culturally relevant knowledge, support, and resources is needed for local dementia caregivers, especially seeing the current Covid-19 outbreak and the new normal in the future.

Primary Objective The current study aims to design and develop a mobile-based multi-component intervention (i.e. an app) to promote mental health among informal caregivers of individuals with dementia in Singapore, and pilot-test the effectiveness of the app among a convenience sample of local informal dementia caregivers.

Secondary Objective(s) Secondary objectives include 1) seeking users' feedback and identifying areas for future improvements; 2) exploring the potential for future bigger trials; 3) providing a development framework for future similar programs.

ELIGIBILITY:
Inclusion Criteria:

1. aged 21 or above;
2. Singapore citizen or permanent resident;
3. primary caregiver who is currently taking care of a PWD;
4. scores 4 and above using the 4-item screening version Zarit Burden Interview;
5. has sufficient skills in using mobile apps;
6. able to read, write, and speak in English

Exclusion Criteria:

1. Caregivers who are pregnant
2. caregivers with vision and hearing problems

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Baseline depressive symptom | baseline - before the intervention
  Centre for Epidemiological Study Scale (0-60), with a higher score indicating a more severe depressive symptom
Post-intervention depressive symptom | within 2 weeks after the intervention
  Centre for Epidemiological Study Scale (0-60), with a higher score indicating a more severe depressive symptom

SECONDARY OUTCOMES:
Baseline knowledge of dementia | baseline - before the intervention
  Dementia Knowledge Assessment Scale (0-54), with higher score indicating better knowledge on dementia
Post intervention knowledge of dementia | within 2 weeks after the intervention
  Dementia Knowledge Assessment Scale (0-54), with higher score indicating better knowledge on dementia
Baseline caregiving self-efficacy | baseline - before the intervention
  Revised Scale for Caregiving Self-efficacy (0-100), with higher score indicating more confidence in caregiving
Post intervention caregiving self-efficacy | within 2 weeks after the intervention
  Revised Scale for Caregiving Self-efficacy (0-100), with higher score indicating more confidence in caregiving
Baseline coping strategy | baseline - before the intervention
  brief Coping Orientation to Problems Experienced inventory - it has a total of 14 subscales, for each subscale higher score indicating more frequent usage of that specific coping strategy
Post intervention coping strategy | within 2 weeks after the intervention
  brief Coping Orientation to Problems Experienced inventory - it has a total of 14 subscales, for each subscale higher score indicating more frequent usage of that specific coping strategy
Baseline positive aspects of caregiving | baseline - before the intervention
  Positive Aspects of Caregiving Scale (9-45) - with a higher score indicates a more positive caregiving experience
Post intervention positive aspects of caregiving | within 2 weeks after the intervention
  Positive Aspects of Caregiving Scale (9-45) - with a higher score indicates a more positive caregiving experience
Baseline caregiver burden | baseline - before the intervention
  Zarit burden interview (0-88) - with a higher score indicating higher perceived caregiving burden
Post intervention caregiver burden | within 2 weeks after the intervention
  Zarit burden interview (0-88) - with a higher score indicating higher perceived caregiving burden
Baseline anxiety level | baseline - before the intervention
  Generalized Anxiety Disorder 7-item scale (0-21) - with a higher score indicating higher anxiety level
Post intervention anxiety level | within 2 weeks after the intervention
  Generalized Anxiety Disorder 7-item scale (0-21) - with a higher score indicating higher anxiety level
Baseline mental well-being | baseline - before the intervention
  Short Positive Mental Health instrument (1-6) - with a higher score indicating higher positive mental health
Post intervention mental well-being | within 2 weeks after the intervention
  Short Positive Mental Health instrument (1-6) - with a higher score indicating higher positive mental health

CONTACTS AND LOCATIONS:
Overall Officials: Qi Yuan, PhD, Principal Investigator — Research Division, Institute of Mental Health
Locations (1):
- Clinic B, Institute of Mental Health, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Our IRB requires a signed research collaboration agreement before we can share the data. Parties who are interested in the current study can write in to inquire about the procedures.

REFERENCES:
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Brown EL, Ruggiano N, Page TF, Roberts L, Hristidis V, Whiteman KL, Castro J. CareHeroes Web and Android Apps for Dementia Caregivers: A Feasibility Study. Res Gerontol Nurs. 2016 Jul-Aug;9(4):193-203. doi: 10.3928/19404921-20160229-02. Epub 2016 Mar 4. PMID 29977440
- [Background] Callan JA, Siegle GJ, Abebe K, Black B, Martire L, Schulz R, Reynolds C 3rd, Hall MH. Feasibility of a pocket-PC based cognitive control intervention in dementia spousal caregivers. Aging Ment Health. 2016;20(6):575-82. doi: 10.1080/13607863.2015.1031635. Epub 2015 May 6. PMID 25945597
- [Background] Fogg, B. J. (2009). A behavior model for persuasive design. Paper presented at the Proceedings of the 4th international Conference on Persuasive Technology.
- [Background] Lorca-Cabrera J, Grau C, Marti-Arques R, Raigal-Aran L, Falco-Pegueroles A, Albacar-Rioboo N. Effectiveness of health web-based and mobile app-based interventions designed to improve informal caregiver's well-being and quality of life: A systematic review. Int J Med Inform. 2020 Feb;134:104003. doi: 10.1016/j.ijmedinf.2019.104003. Epub 2019 Nov 23. PMID 31790857
- [Background] McCurdie T, Taneva S, Casselman M, Yeung M, McDaniel C, Ho W, Cafazzo J. mHealth consumer apps: the case for user-centered design. Biomed Instrum Technol. 2012 Fall;Suppl:49-56. doi: 10.2345/0899-8205-46.s2.49. No abstract available. PMID 23039777
- [Background] Rathnayake S, Moyle W, Jones C, Calleja P. mHealth applications as an educational and supportive resource for family carers of people with dementia: An integrative review. Dementia (London). 2019 Oct-Nov;18(7-8):3091-3112. doi: 10.1177/1471301218768903. Epub 2018 Apr 9. No abstract available. PMID 29631492
- [Background] Reyes, A. K., Camargo, J. E., & Díaz, G. M. (2015). Design of a mobile application to support non-pharmacological therapies for people with Alzheimer disease. Paper presented at the International Conference on Smart Health.
- [Background] Sallim AB, Sayampanathan AA, Cuttilan A, Ho R. Prevalence of Mental Health Disorders Among Caregivers of Patients With Alzheimer Disease. J Am Med Dir Assoc. 2015 Dec;16(12):1034-41. doi: 10.1016/j.jamda.2015.09.007. PMID 26593303
- [Background] Sikder AT, Yang FC, Schafer R, Dowling GA, Traeger L, Jain FA. Mentalizing Imagery Therapy Mobile App to Enhance the Mood of Family Dementia Caregivers: Feasibility and Limited Efficacy Testing. JMIR Aging. 2019 Mar 21;2(1):e12850. doi: 10.2196/12850. PMID 31518275
- [Background] Subramaniam M, Chong SA, Vaingankar JA, Abdin E, Chua BY, Chua HC, Eng GK, Heng D, Hia SB, Huang W, Jeyagurunathana A, Kua J, Lee SP, Mahendran R, Magadi H, Malladi S, McCrone P, Pang S, Picco L, Sagayadevan V, Sambasivam R, Seng KH, Seow E, Shafie S, Shahwan S, Tan LL, Yap M, Zhang Y, Ng LL, Prince M. Prevalence of Dementia in People Aged 60 Years and Above: Results from the WiSE Study. J Alzheimers Dis. 2015;45(4):1127-38. doi: 10.3233/JAD-142769. PMID 25672767
- [Background] Yuan Q, Wang P, Tan TH, Devi F, Poremski D, Magadi H, Goveas R, Ng LL, Chong SA, Subramaniam M. Coping Patterns Among Primary Informal Dementia Caregivers in Singapore and Its Impact on Caregivers-Implications of a Latent Class Analysis. Gerontologist. 2021 Jul 13;61(5):680-692. doi: 10.1093/geront/gnaa080. PMID 32592582
- [Derived] Yuan Q, Lee YT, Samari E, Zhang Y, Goveas R, Ng LL, Subramaniam M. Evaluating the feasibility and potential effectiveness of a mobile-based intervention to promote the mental health of informal caregivers of persons with dementia in Singapore: Results from a mixed-methods two-arm pilot randomized controlled trial. J Affect Disord. 2026 Apr 15;399:121059. doi: 10.1016/j.jad.2025.121059. Epub 2025 Dec 29. PMID 41475574
- [Derived] Lee YT, Yuan Q, Zhang Y, Samari E, Goveas R, Ng LL, Subramaniam M. Evaluating a mobile-based intervention to promote the mental health of informal dementia caregivers in Singapore: Study protocol for a pilot two-armed randomised controlled trial. PLoS One. 2024 Jun 24;19(6):e0305729. doi: 10.1371/journal.pone.0305729. eCollection 2024. PMID 38913625
- See also: World Alzheimer Report 2015, The Global Impact of Dementia: An Analysis of Prevalence, Incidence, Cost and Trends — https://www.alz.co.uk/research/WorldAlzheimerReport2015.pdf
- See also: ANNUAL SURVEY ON INFOCOMM USAGE IN HOUSEHOLDS AND BY INDIVIDUALS FOR 2017 — https://www.imda.gov.sg/-/media/imda/files/industry-development/fact-and-figures/infocomm-survey-reports/hh2017-survey.pdf?la=en